CLINICAL TRIAL: NCT02155491
Title: Global Anticoagulant Registry in the Field Observing Treatment and Outcomes in Patients With Treated Acute Venous Thromboembolic Events in the Real World
Brief Title: Global Anticoagulant Registry in the FIELD- Venous Thromboembolic Events
Acronym: GARFIELD-VTE
Status: Completed | Type: Observational
Sponsor: Thrombosis Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: TRI08889
Record Dates: First submitted 2014-04-30; First posted 2014-06-04 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: venous, thromboembolism, embolism, DVT, Pulmonary Embolism, thrombosis
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Thromboembolism; Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective cohort 1: In order to observe temporal trends in management of VTE a first cohort of 5000 consecutive unselected patients treated for acute VTE will be recruited. This cohort will take approximately 9 months to recruit. Potential patients must be assessed for eligibility within 30 days of their acute VTE diagnosis. They will be followed prospectively for 36 months.
- Prospective cohort 2: In order to observe temporal trends in management of VTE a second cohort of 5000 consecutive unselected patients treated for acute VTE will be recruited. Recruitment into the second cohort will commence when recruitment is completed in the first cohort. This cohort will take approximately 9 months to recruit. Potential patients must be assessed for eligibility within 30 days of their acute VTE diagnosis. They will be followed prospectively for 36 months.

SUMMARY:
The protocol is a large registry to describe acute, sub-acute and extended duration of anticoagulation management, clinical and economic duration of anticoagulation management, clinical and economic outcomes in patients with treated acute VTE (DVT and PE) in the real-world setting.

Main objectives are to clarify the:

* treatment related details for acute VTE (either conventional anticoagulation therapy, treatment with a direct oral anti-coagulant or other modalities of treatment)
* Rate of early and late symptomatic VTE recurrence
* Rate and nature of complications of VTE including post thrombotic syndrome and chronic thromboembolic pulmonary hypertension
* Rate of bleeding complications
* Rate of all-cause mortality at six months

DETAILED DESCRIPTION:
Other objectives are to clarify the additional outcomes of:

* Stroke (Measured by number of incidences)
* Transient Ischemic Attack (TIA) (Measured by number on incidences)
* ST Elevated Myocardial Infarction (STEMI) (Measured by number of incidences)
* Non-ST Elevated Myocardial Infraction (NSTEMI) (Measured by number of incidences)
* Unstable Angina (Measured by number of incidences)
* Quality of life and patient reported outcomes and costs associated with the management of VTE.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years and over
* Treated first time or recurrent DVT (lower or upper extremity), PE alone or overlapping DVT and PE confirmed by appropriate diagnostic methods (patients must be assessed for eligibility within 30 days of diagnosis)
* Patients included with recurrent VTE must have completed treatment for the previous VTE episode

Exclusion Criteria:

* Patients for whom long-term follow-up is not envisaged within the enrolling hospital or the associated primary care physician
* Patients participating in an interventional study that dictates treatments, visit frequency, or diagnostic procedures
* Patients with only superficial vein thrombosis (SVT)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sites will be selected at random from a representative list reflecting treatment patterns in each country. Consecutive male and female VTE patients at the randomly selected sited will be included in the registry if they meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10679 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of recurrent symptomatic VTE (DVT and fatal or non-fatal PE) | 36 months
  Rate of recurrent symptomatic VTE (DVT and fatal or non-fatal PE)
Bleeding events | 36 months
  Frequency, location, severity (classified as major or non-major)
Hospitalization | 36 months
  Measured by number of occurrences.
Post Thrombotic Syndrome | 36 months
  Measured by number of occurrences and severity.
Chronic thromboembolic pulmonary hypertension | 36 months
  Measured by number of occurrences and severity.
IVC filter placement | 36 months
  Measured by number of occurrences.
Other urgent interventions for VTE | 36 months
  Measured by number of occurrences.
Anticoagulation therapy persistence | 36 months
  Estimation of Anticoagulation therapy will be compared to actual total time Anticoagulation therapy was used by patients.
All cause of mortality | 36 months
  Causes of death: PE, stroke, cardiac, cancer-related, other...
International Normalized Ratio (INR) Values in Patients treated with Vitamin K Antagonists | 36 months
  Will be assessed by frequency of INR monitoring, and number of INR readings taken before patient achieved optimum range.

SECONDARY OUTCOMES:
Stroke | 36 months
  Ischemic stroke, hemorrhagic stroke
Trans Ischemic Attack (TIA) | 36 months
  Measured by number of occurrences.
Myocardial Infarction | 36 months
  Measured by number of occurrences of both ST-Elevated Myocardial Infarction and Non-ST Elevated Myocardial Infarction (STEMI/NSTEMI).
Unstable angina | 36 months
  Measured by number of occurrences.
Quality of life and patient treatment satisfaction over a three year period | 36 months
  Measured by Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K Kakkar, MD, Study Director — Thrombosis Research Institute
Locations (1):
- Dr Terence Hart, Muscle Shoals, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heit JA. The epidemiology of venous thromboembolism in the community. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):370-2. doi: 10.1161/ATVBAHA.108.162545. No abstract available. PMID 18296591
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] Eurostat, Eurostat statistics on health and safety 2001.
- [Background] Silverstein MD, Heit JA, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Trends in the incidence of deep vein thrombosis and pulmonary embolism: a 25-year population-based study. Arch Intern Med. 1998 Mar 23;158(6):585-93. doi: 10.1001/archinte.158.6.585. PMID 9521222
- [Background] Prandoni P, Noventa F, Ghirarduzzi A, Pengo V, Bernardi E, Pesavento R, Iotti M, Tormene D, Simioni P, Pagnan A. The risk of recurrent venous thromboembolism after discontinuing anticoagulation in patients with acute proximal deep vein thrombosis or pulmonary embolism. A prospective cohort study in 1,626 patients. Haematologica. 2007 Feb;92(2):199-205. doi: 10.3324/haematol.10516. PMID 17296569
- [Background] Kahn SR, Ginsberg JS. Relationship between deep venous thrombosis and the postthrombotic syndrome. Arch Intern Med. 2004 Jan 12;164(1):17-26. doi: 10.1001/archinte.164.1.17. PMID 14718318
- [Background] Prandoni P, Kahn SR. Post-thrombotic syndrome: prevalence, prognostication and need for progress. Br J Haematol. 2009 May;145(3):286-95. doi: 10.1111/j.1365-2141.2009.07601.x. Epub 2009 Feb 13. PMID 19222476
- [Background] Leizorovicz A. Long-term consequences of deep vein thrombosis. Haemostasis. 1998;28 Suppl 3:1-7. doi: 10.1159/000022399. PMID 10069756
- [Background] Prandoni P, Lensing AW, Prins MR. Long-term outcomes after deep venous thrombosis of the lower extremities. Vasc Med. 1998;3(1):57-60. doi: 10.1177/1358836X9800300112. PMID 9666534
- [Background] Ruppert A, Steinle T, Lees M. Economic burden of venous thromboembolism: a systematic review. J Med Econ. 2011;14(1):65-74. doi: 10.3111/13696998.2010.546465. Epub 2011 Jan 12. PMID 21222564
- [Background] MacDougall DA, Feliu AL, Boccuzzi SJ, Lin J. Economic burden of deep-vein thrombosis, pulmonary embolism, and post-thrombotic syndrome. Am J Health Syst Pharm. 2006 Oct 15;63(20 Suppl 6):S5-15. doi: 10.2146/ajhp060388. PMID 17032933
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Hyers TM, Agnelli G, Hull RD, Morris TA, Samama M, Tapson V, Weg JG. Antithrombotic therapy for venous thromboembolic disease. Chest. 2001 Jan;119(1 Suppl):176S-193S. doi: 10.1378/chest.119.1_suppl.176s. No abstract available. PMID 11157648
- [Background] McRae SJ, Ginsberg JS. Initial treatment of venous thromboembolism. Circulation. 2004 Aug 31;110(9 Suppl 1):I3-9. doi: 10.1161/01.CIR.0000140904.52752.0c. PMID 15339875
- [Background] Kearon C, Akl EA, Comerota AJ, Prandoni P, Bounameaux H, Goldhaber SZ, Nelson ME, Wells PS, Gould MK, Dentali F, Crowther M, Kahn SR. Antithrombotic therapy for VTE disease: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e419S-e496S. doi: 10.1378/chest.11-2301. PMID 22315268
- [Background] Adcock, D.M., Recurrence of thromboembolism: determining risk. Clinical Haemostasis Review. 2005. 19:1.
- [Background] Spyropoulos AC, Lin J. Direct medical costs of venous thromboembolism and subsequent hospital readmission rates: an administrative claims analysis from 30 managed care organizations. J Manag Care Pharm. 2007 Jul-Aug;13(6):475-86. doi: 10.18553/jmcp.2007.13.6.475. PMID 17672809
- [Background] Summary of Recommendation Statements. Kidney Int Suppl (2011). 2013 Jan;3(1):5-14. doi: 10.1038/kisup.2012.77. No abstract available. PMID 25598998
- [Derived] Goto S, Turpie AGG, Farjat AE, Weitz JI, Haas S, Ageno W, Goldhaber SZ, Angchaisuksiri P, Kayani G, MacCallum P, Schellong S, Bounameaux H, Mantovani LG, Prandoni P, Kakkar AK; GARFIELD-VTE investigators. The influence of anemia on clinical outcomes in venous thromboembolism: Results from GARFIELD-VTE. Thromb Res. 2021 Jul;203:155-162. doi: 10.1016/j.thromres.2021.05.007. Epub 2021 May 15. PMID 34023735
- [Derived] Weitz JI, Haas S, Ageno W, Goldhaber SZ, Turpie AGG, Goto S, Angchaisuksiri P, Nielsen JD, Kayani G, Farjat AE, Schellong S, Bounameaux H, Mantovani LG, Prandoni P, Kakkar AK; GARFIELD-VTE investigators. Cancer associated thrombosis in everyday practice: perspectives from GARFIELD-VTE. J Thromb Thrombolysis. 2020 Aug;50(2):267-277. doi: 10.1007/s11239-020-02180-x. PMID 32583306
- See also: Global Anticoagulant Registry in the FIELD, Venous thromboembolism Event (GARFIELD-VTE) — http://www.tri-london.ac.uk/garfield-vte